CLINICAL TRIAL: NCT07275749
Title: The Safety and Efficacy of Acetyl-leucine in Post-stroke Ataxia: a Randomized Placebo-controlled Trial
Brief Title: Acetyl-leucine in Post-stroke Ataxia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed G. zeinhom, MD, Dr, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19012025
Record Dates: First submitted 2025-11-24; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Stroke
Keywords: Acetyl-leucine; post-stroke ataxia; posterior-circulation stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Clopidogrel; Tablets; Aspirin

STUDY DESIGN:
Intervention Model Description: the investigators will conduct our double-blinded, placebo-controlled, parallel-group trial in Kafr-Elsheikh University in the time between 1st January 2026 to 1st July 2026.
  Our study will include 200 post-circulation AIS patients who will undergo randomization and divided into two groups; The (A) group, which consisted of 100 patients who administered (a 4 gram of acetyl-leucine per day) and the (B) group, which had 100 patients who administered a placebo during the first 24 hours of stroke onset and for 3 months.
  Both groups received (open-label 300 mg loading dose aspirin and 300 mg loading clopidogrel during the first 24 hours of stroke onset, followed by 75 mg clopidogrel and 100 mg aspirin once daily from the 2nd to the 90th day.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An independent statistician generated a blocked randomisation sequence using computer-generated random numbers; in a one-to-one ratio, participants were randomly assigned to receive a 4 gram of acetyl-leucine per day or placebo by a specially trained and qualified nurse.
  We prepared Sequentially numbered 200 labels for each Drug A or B. According to the randomisation chart. Envelopes were attached to the patient's files. Patients were recruited sequentially and were given enrolment numbers starting from 1, which were mentioned in their files. Files with the same number as the patient enrolment number were opened, and the patients were assigned to receive drugs A or B. Drug A included acetyl-leucine , and Drug B included placebo. Both groups received an open-label 300 mg loading dose aspirin and 300 mg loading clopidogrel during the first 24 hours of stroke onset, followed by 75 mg clopidogrel and 100 mg aspirin once daily from the 2nd to the 90th day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- acetyl-leucine (Active Comparator): The acetyl-leucine arm will receive (a 4 gram of acetyl-leucine daily for three months and an open-label loading 300 mg aspirin and 300 mg clopidogrel during the first 24 hours of stroke, followed by a maintenance dose of 100 mg aspirin and 75 mg clopidogrel.
  Interventions: Drug: Acetyl-Leucine; Drug: Clopidogrel 75 Mg Oral Tablet; Drug: aspirin 100mg
- placebo (Placebo Comparator): The placebo arm will receive 4 gram placebo daily for three months and an open-label loading 300 mg aspirin and 300 mg clopidogrel during the first 24 hours of stroke, followed by a maintenance dose of 100 mg aspirin and 75 mg clopidogrel.
  Interventions: Drug: Placebo; Drug: Clopidogrel 75 Mg Oral Tablet; Drug: aspirin 100mg

INTERVENTIONS:
Drug: Acetyl-Leucine — The acetyl-leucine arm will receive (a 4 gram of acetyl-leucine daily for three months and an open-label loading 300 mg aspirin and 300 mg clopidogrel during the first 24 hours of stroke, followed by a maintenance dose of 100 mg aspirin and 75 mg clopidogrel.
  Other Names: group A
  Arms: acetyl-leucine
Drug: Placebo — The placebo arm will receive (a 4 gram of placebo daily for three months and an open-label loading 300 mg aspirin and 300 mg clopidogrel during the first 24 hours of stroke, followed by a maintenance dose of 100 mg aspirin and 75 mg clopidogrel.
  Arms: placebo
Drug: Clopidogrel 75 Mg Oral Tablet — All patients received an open-label loading 300 mg clopidogrel during the first 24 hours of stroke, followed by a maintenance dose of 75 mg clopidogrel once daily.
Drug: aspirin 100mg — All patients received an open-label loading 300 mg aspirin during the first 24 hours of stroke, followed by a maintenance dose of 100 mg aspirin once daily.

SUMMARY:
Along with the current clinical trial, the efficacy and safety of 4 gram of acetyl-leucine daily for three months in patients with post-stroke ataxia following posterior-circulation ischaemic stroke assessed through BBS, SARA, and mRS, and possible adverse effects.

DETAILED DESCRIPTION:
the investigators will conduct our double-blinded, placebo-controlled, parallel-group trial in Kafr-Elsheikh University in the time between 1st January 2026 to 1st July 2026.

the study will include 200 post-circulation AIS patients who will undergo randomization and divided into two groups; The (A) group, which consisted of 100 patients who administered (a 4 gram of acetyl-leucine per day) and the (B) group, which had 100 patients who administered a placebo during the first 24 hours of stroke onset and for 3 months.

Both groups received (open-label 300 mg loading dose aspirin and 300 mg loading clopidogrel during the first 24 hours of stroke onset, followed by 75 mg clopidogrel and 100 mg aspirin once daily from the 2nd to the 90th day.

The diagnosis of ischemic stroke was established through a detailed clinical history and examination and suitable brain imaging. All of the patients had CT of the brain and CT angiography (CTA) including the aortic arch through the circle of Willis before thrombolysis; the CT of the brain was performed on the 64-slice dual-source spiral CT scanner of Somatom definition by Siemens, and the supratentorial compartment scans were imaged with 5-8mm contiguous sections and the brain stem and cerebellum scans were imaged with 3-5mm slices, and we obtained eighteen images for each series. After thrombolysis, all of the patients underwent an MRI brain on a 1.5 T (Siemens Essenza) MR system, stroke protocol: T1W, T2W, fluid attenuation inversion recovery imaging (FLAIR), diffusion-weighted imaging (DWI), T2 Echo Gradient, and MRA brain & neck time of flight (TOF) if CTA was contraindicated; the investigators performed an additional brain CT scan after 24-36 hours to evaluate hemorrhagic transformation. (8), and considered hemorrhagic transformation symptomatic if the NIHSS score increased by 4 points or more. (9) The computed tomography (CT)/ magnetic resonance imaging (MRI) examinations were assessed in our study by two highly experienced professionals: a senior stroke physician and a senior radiologist.

the investigators identified posterior-circulation stroke (PCS) when ischemic occlusion affected basilar, posterior cerebral or vertebral arteries

ELIGIBILITY:
Inclusion Criteria:

* the investigators included both males and females, aged between 18 and 80 years, who experienced their first-ever posterior-circulation ischaemic stroke and presented with gait ataxia and score at least 1 point on the items gait, stance, trunk or heel-shin-slide of the Scale for the Assessment and Rating of Ataxia (SARA) and 47 points or less on the Berg Balance Scale (BBS).
* All of our patients underwent randomisation during the first 24 hours of the symptoms' onset, and within the first 24 hours from the time at which the patient's condition was last reported to be normal for wake-up stroke patients.

Exclusion Criteria:

* the investigators excluded patients with modified Rankin Scale (mRS) score of 5 or more, physical or mental conditions that would not allow safe participation in the study or would influence the assessment of outcomes (e.g., dementia, disturbed conscious level, severe aphasia, etc.).
* the investigators ruled out participants who suffered from neurological diseases associated with recurrent neurological deficits, such as (epilepsy, multiple sclerosis, head trauma followed by neurological deficit).
* the investigators excluded participants who underwent intravenous thrombolysis, carotid, cerebrovascular, or coronary revascularization during the first week of the trial to avoid clouding of efficacy and safety analysis.
* the investigators excluded patients who experienced recurrent ischemic stroke detected from their clinical data and/or magnetic resonance imaging (MRI) brain findings. In addition, we excluded participants who experienced hypersensitivity to the study treatment
* the investigators excluded participants who experienced organ failure such as renal failure and liver cell failure, active malignancies, and patients with a known bleeding diathesis or coagulation disorder, a history of intracerebral hemorrhage, gastrointestinal bleeding within the past 6 months, or major surgery within 30 days before randomisation .

the investigators excluded pregnant and lactating women, patients with cerebral venous thrombosis, and patients with stroke associated with cardiac arrest.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
value of the Berg balance scale (BBS) | 90 days
  the primary efficacy endpoint is balance as assessed using the BBS (14). The BBS is considered the gold standard for evaluating balance in people after stroke (20).
  a 14-item test that assesses an individual's balance and risk of falling. It measures static and dynamic balance through a series of tasks, with each item scored on a scale of 0 to 4, for a total possible score of 56, with higher score related to more impairment in balance
the rate of participants who suffered from treatment-related side effects | 90 days
  the primary safety endpoint the rate of participants who suffered from treatment-related side effects assessed via questionnaire.

SECONDARY OUTCOMES:
value of Scale for the Assessment and Rating of Ataxia (SARA) | 90 days
  the first secondary efficacy endpoint is the severity of ataxic symptoms, as determined by the Scale for the Assessment and Rating of Ataxia (SARA)
  The SARA is a tool for assessing ataxia. It has eight categories with accumulative score ranging from 0 (no ataxia) to 40 (most severe ataxia).
value of Modified Rankin Scale(mRS) at three months | 90 days
  mRS Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability; its value ranges from 0 to 6; the lower the score, the better the stroke outcome. A favourable stroke outcome is considered with mRS value equal to two or less.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed G. Zeinhom, MD, Study Director — neurology department kafr el-sheikh university
Locations (1):
- Kafr Elsheikh University Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No
All the data that support the findings of this research will be available from the corresponding author M. Zeinhom upon reasonable request.

REFERENCES:
- [Result] Paciaroni M, Ince B, Hu B, Jeng JS, Kutluk K, Liu L, Lou M, Parfenov V, Wong KSL, Zamani B, Paek D, Min Han J, Del Aguila M, Girotra S. Benefits and Risks of Clopidogrel vs. Aspirin Monotherapy after Recent Ischemic Stroke: A Systematic Review and Meta-Analysis. Cardiovasc Ther. 2019 Dec 1;2019:1607181. doi: 10.1155/2019/1607181. eCollection 2019. PMID 31867054
- [Result] Lipton RB, Liberman JN, Kolodner KB, Bigal ME, Dowson A, Stewart WF. Migraine headache disability and health-related quality-of-life: a population-based case-control study from England. Cephalalgia. 2003 Jul;23(6):441-50. doi: 10.1046/j.1468-2982.2003.00546.x. PMID 12807523